CLINICAL TRIAL: NCT04759040
Title: Migraineguard ™ Supplement Reduces the Severity and Frequency of Migraine , a Randomized, Placebo-controlled, Double-blind, Trial
Brief Title: Improvement of Migraine Severity and Frequency With Migraineguard ™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbacure Natural (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MIGRAINEGUARD
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Migraine; Headache
Keywords: migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MigraineGuard (Active Comparator): Active supplement treatment , MigraineGuard capsule containing Coq10 , Magnesium ,Vit B2 , Skullcap Extract , Feverfew Extract , Piperine
  Interventions: Dietary Supplement: Migraineguard
- Placebo for MigraineGuard (Placebo Comparator): Placebo capsules non identifiable from Migraineguard capsules were used as control comparator
  Interventions: Dietary Supplement: Migraineguard

INTERVENTIONS:
Dietary Supplement: Migraineguard — 2 Capsules per day for 7 Months

SUMMARY:
Numerous treatments have been recommended for the prevention of migraine. The purpose of this randomized double-blind placebo controlled trial was to assess the efficacy of MIGRAINEGUARD ™ supplement by Herbacure Natural containing a combination of COQ10 , magnesium, riboflavin ,feverfew , Skullcap and black pepper as prophylactic treatment for migraine.

DETAILED DESCRIPTION:
Our team will assess MIGRAINEGUARD ™ , a migraine prevention supplement marketed Herbacure Natural for individual suffering from multiple migraine attacks in one month . The purpose of this 7-months , randomized, double-blind, placebo controlled study is to evaluate the efficacy and safety of MIGRAINEGUARD ™ produced by Herbacure Natural , A Canadian company based in Vancouver , BC , in reducing migraine headache severity and frequency of attacks compared to placebo when used every day, as a preventative solution for migraine and to assess and monitor the safety of its usage for adverse effects.

The primary end-point is the severity and the frequency reduction of migraine attacks. The secondary end-points will be the existence of adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 to 65 years Female and Male
* Based on IHS criteria ,are diagnosed with migraine (criteria of the International Classification of Headaches Disorders)
* Individuals with minimum of 3 severe to extreme migraine attacks during the last 3 months .
* Generally in good health

Exclusion Criteria:

* Individuals taking any preventive treatment for migraine
* Excessive usage of painkillers
* Cancer & Head injury and trauma
* Any medical condition that may impact the validity of collected information
* Previous usage of Botox within 6 months of study
* Last week usage of triptans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Number of patient experiencing migraine attack reduction by at least 50 percent in one month . | 7 months
  Number of patient experiencing migraine attack reduction by at least 50 percent in one month . Migraineurs with 50 percent migraine attack decrease are considered "Responders" to supplement.
Severity of migraine headache reduction after & Months | 7 Months
  Reduction of Migraine severity After 7 months of supplementation

SECONDARY OUTCOMES:
Adverse Reactions | 7 months
  Report of any adverse reaction due to supplementation during the study

CONTACTS AND LOCATIONS:
Overall Officials: AMIR A DOWLATSHAHI, PHD, Study Director — HERBACURE NATURAL INC
Locations (1):
- Herbacure Natural, Burnaby, British Columbia, Canada